CLINICAL TRIAL: NCT00922350
Title: Heliox and Posture Optimize Action of Nebulization With Bronchodilators for Asthma Attacks. Randomized Trial.
Brief Title: Heliox and Posture in Patients With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Daniella Cunha Brandão, Department of Physiotherapy
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2525
Record Dates: First submitted 2009-06-08; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Acute Asthma
Keywords: asthma; heliox; bronchodilators; posture
MeSH Terms: conditions — Asthma | interventions — heliox; MUSK protein, human; Oxygen; NPSR1 protein, human; Posture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- heliox (Experimental): The patients in this group underwent nebulization with heliox carried by the trunk erect
  Interventions: Other: HELIOX
- heliox+posture (Experimental): The patients in this group carried out the mist carried by heliox and the trunk tilted forward
  Interventions: Other: HELIOX+POSTURE
- oxygen+posture (Experimental): The patients in this group carried out the mist carried by oxygen and the trunk tilted forward
  Interventions: Other: OXYGEN + POSTURE
- oxygen (Active Comparator): The patients in this group carried out the mist carried by the oxygen and the trunk upright
  Interventions: Other: OXYGEN

INTERVENTIONS:
Other: HELIOX — The nebulization was conducted in the same way that heliox + posture group, except the attitude of trunk, where the patients in this group did the Nebulizer with the trunk upright.
  Other Names: asma
  Arms: heliox
Other: OXYGEN — The NEBULIZATION was performed the same way as the heliox group, except for torso posture, where the patients in this group with the trunk upright Nebulizer Oxygen for cars have A NEBULIZATION.
  Other Names: ASTHMA; NEBULIZATION
  Arms: oxygen
Other: HELIOX+POSTURE — Patients underwent two carried by heliox nebulization associated with fenoterol (2.5 mg) and ipratropium bromide (0.25 mg). We used three ml of saline solution at 0.9%. For nebulization with heliox or oxygen, was used a system of distribution not invasive, semi-closed in a mask that is non toxic connected to a piece "Y" with a nebulizer in a follow and a bag of tank with a capacity for 2.5 L in the other connected with a valve action. This system was used so that there was a dilution gas. The proportion of 80:20 heliox was used (80% helium: 20% oxygen). To postural change in groups and heliox Oxygen + posture + posture, oriented to the participants to maintain an angle of inclination of the trunk and elbows supported on the thighs, measured from the anterior axillary line and lateral epicondyle of the femur, between 50th and 60th .
  Other Names: heliox; posture; physioterapy
  Arms: heliox+posture
Other: OXYGEN + POSTURE — The NEBULIZATION was conducted in the same way that heliox + posture GROUP, however the patients in this group have the Oxygen for Carr A NEBULIZATION
  Other Names: POSTURE; PHYSIOTERAPY; ASTHMA
  Arms: oxygen+posture

SUMMARY:
The purpose of this study is to verify that nebulization with bronchodilators associated with heliox gas (helium + oxygen) and the posture of a leaning forward truck is effective in patients with an asthma attack.

DETAILED DESCRIPTION:
When associated with inhaled bronchodilators, the heliox, a mixture of helium and oxygen in obstructive lung diseases with asthma, reduces the turbulence of airflow despite high rates, due to its low density.

Although the first report of the use of heliox in the treatment of asthma dating to 1935, few controlled studies are available clarify the impact of the use of heliox in hospital admission of patients with acute asthma attacks refractory to standard treatment.

The severe airflow obstruction, observed in cases of acute asthma, also leads to lung hyperinflation that favors the increase of respiratory work by increasing the load for the inspiratory muscles by placing them at a mechanical disadvantage.

Various body positions were studied relating them to muscle activity with mechanical disadvantage. These studies suggest that the influence posture acts mainly in the position of the diaphragm, thus, increasing the stress related to other muscles such as the abdominals and the effect of gravity on these.

This study aims to: assess the efficiency of the positioning body associated with nebulization with bronchodilators carried by heliox during acute severe asthma in adults, using as the primary outcomes FEV1, FVC and PEF and secondary outcomes as the Borg scale, inspiratory capacity, RR, HR and SpO2.

ELIGIBILITY:
Inclusion Criteria:

* reversibility of bronchial obstruction after administration of bronchodilator drugs for at least 10% in FEV1
* a clinical diagnosis of acute severe asthma
* a history of asthma over 1 year
* duration of the crisis of current asthma lasting less than seven days

Exclusion Criteria:

* were unable to understand or perform the spirometric maneuver
* smoking (within the last 3 years associated with a higher consumption of 100 cigarettes/year)
* other pulmonary comorbidities
* lower to upper airways
* heart failure
* heart rate greater than 150 bpm
* systolic pressure below 90 mmHg or greater than 150 MHG
* pregnancy
* inability to stay inline with the trunk forward

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Spirometry | 6 months

SECONDARY OUTCOMES:
Respiratory rate | 6 months
Peripheral oxygen saturation | 6 months
Borg scale | 6 months
Heart rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Armele Andrade, Study Director — Universidade Federal de Pernambuco
Locations (1):
- Barros Lima Policlinic, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Kass JE, Terregino CA. The effect of heliox in acute severe asthma: a randomized controlled trial. Chest. 1999 Aug;116(2):296-300. doi: 10.1378/chest.116.2.296. PMID 10453854
- [Result] Hess DR, Fink JB, Venkataraman ST, Kim IK, Myers TR, Tano BD. The history and physics of heliox. Respir Care. 2006 Jun;51(6):608-12. PMID 16723037
- [Result] Hess DR, Acosta FL, Ritz RH, Kacmarek RM, Camargo CA Jr. The effect of heliox on nebulizer function using a beta-agonist bronchodilator. Chest. 1999 Jan;115(1):184-9. doi: 10.1378/chest.115.1.184. PMID 9925082
- [Result] Gorini M, Iandelli I, Misuri G, Bertoli F, Filippelli M, Mancini M, Duranti R, Gigliotti F, Scano G. Chest wall hyperinflation during acute bronchoconstriction in asthma. Am J Respir Crit Care Med. 1999 Sep;160(3):808-16. doi: 10.1164/ajrccm.160.3.9712088. PMID 10471601
- [Derived] Brandao DC, Britto MC, Pessoa MF, de Sa RB, Alcoforado L, Matos LO, Silva TN, de Andrade AD. Heliox and forward-leaning posture improve the efficacy of nebulized bronchodilator in acute asthma: a randomized trial. Respir Care. 2011 Jul;56(7):947-52. doi: 10.4187/respcare.00963. Epub 2011 Feb 21. PMID 21352660
- See also: Federal University of Pernambuco — http://www.ufpe.br